CLINICAL TRIAL: NCT01815736
Title: A Phase 3, Open-Label Study to Evaluate Switching From a TDF-Containing Combination Regimen to a TAF-Containing Combination Single Tablet Regimen (STR) in Virologically-Suppressed, HIV-1 Positive Subjects
Brief Title: Study to Evaluate Switching From a TDF-Containing Combination Regimen to a TAF-Containing Fixed Dose Combination (FDC) in Virologically-Suppressed, HIV-1 Positive Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-292-0109; 2012-005114-20 (EudraCT Number)
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: HIV; HIV Infections
Keywords: HIV; HIV 1 Infected; Virologically-Suppressed
MeSH Terms: conditions — HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Ritonavir; Atazanavir Sulfate; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- E/C/F/TAF (Experimental): Randomized Phase: Elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) for up to 96 weeks.
  Extension Phase: After completing 96 weeks of randomized treatment, all participants will be given the opportunity to receive open-label E/C/F/TAF until it becomes commercially available, or until Gilead elects to terminate the development of E/C/F/TAF.
  Interventions: Drug: E/C/F/TAF
- Stay on Baseline Treatment Regimen (SBR) (Active Comparator): Randomized Phase: Participants stayed on their baseline emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF)-containing regimen E/C/F/TDF; efavirenz (EFV)/FTC/TDF; ritonavir (RTV)-boosted atazanavir (ATV)+FTC/TDF; or cobicistat (COBI-boosted ATV+FTC/TDF) administered according to prescribing information for up to 96 weeks.
  Extension Phase: After completing 96 weeks of randomized treatment (SBR), all participants will be given the opportunity to receive open-label E/C/F/TAF until it becomes commercially available, or until Gilead elects to terminate the development of E/C/F/TAF.
  Interventions: Drug: E/C/F/TDF; Drug: EFV/FTC/TDF; Drug: RTV; Drug: ATV; Drug: FTC/TDF; Drug: COBI

INTERVENTIONS:
Drug: E/C/F/TAF — 150/150/200/10 mg FDC tablet administered orally once daily
  Other Names: EVG/COBI/FTC/TAF; Genvoya®
  Arms: E/C/F/TAF
Drug: E/C/F/TDF — 150/150/200/300 mg FDC tablet administered orally once daily
  Other Names: Stribild®
  Arms: Stay on Baseline Treatment Regimen (SBR)
Drug: EFV/FTC/TDF — 600/200/300 mg FDC tablet administered orally once daily
  Other Names: Atripla®
  Arms: Stay on Baseline Treatment Regimen (SBR)
Drug: RTV — 100 mg tablet administered orally once daily
  Other Names: Norvir®
  Arms: Stay on Baseline Treatment Regimen (SBR)
Drug: ATV — 300 mg capsule administered orally once daily
  Other Names: Reyataz®
  Arms: Stay on Baseline Treatment Regimen (SBR)
Drug: FTC/TDF — 200/300 mg tablet administered orally once daily
  Other Names: Truvada®
  Arms: Stay on Baseline Treatment Regimen (SBR)
Drug: COBI — 150 mg tablet administered orally once daily
  Other Names: Tybost®; GS-9350
  Arms: Stay on Baseline Treatment Regimen (SBR)

SUMMARY:
The primary objective of this study is to evaluate the non-inferiority of switching to a tenofovir alafenamide (TAF)-containing fixed dose combination (FDC) relative to maintaining tenofovir disoproxil fumarate (TDF)-containing combination regimens in virologically suppressed HIV-infected participants as determined by having HIV-1 RNA < 50 copies/mL at Week 48.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Currently receiving antiretroviral therapy consisting of E/C/F/TDF, EFV/FTC/TDF, RTV+ATV+FTC/TDF, or COBI+ATV+FTC/TDF for ≥ 6 consecutive months preceding the final visit in their earlier study
* Completion of the Week 144 visit in studies GS-US-236-0102, GS-US-236-0103, GS-US-216-0114, or completion of the Week 96 visit in study GS-US-264-0110 (only participants on an EFV-based regimen), or completion of studies GS-US-236-0104, GS-US-216-0105
* Plasma human immunodeficiency virus type 1-ribonucleic acid (HIV-1 RNA) concentrations at undetectable levels for at least 6 consecutive months prior to the screening visit and have HIV RNA < 50 copies/mL at the screening visit
* Normal echocardiograph (ECG)
* Estimated glomerular filtration rate (GFR) ≥ 50 mL/min according to the Cockcroft-Gault formula for creatinine clearance
* Hepatic transaminases (aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) ≤ 5 × upper limit of the normal range (ULN)
* Direct bilirubin ≤ 1.5 x ULN
* Adequate hematologic function
* Serum amylase ≤ 5 × ULN
* Females of childbearing potential must agree to utilize highly effective contraception methods or be non-heterosexually active or practice sexual abstinence from screening throughout the duration of study treatment and for 12 weeks following the last dose of study drug if receiving EFV/FTC/TDF regimen, and 30 days for those assigned to all other regimens.
* Female participants who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing
* Female participants who have stopped menstruating for ≥ 12 months but do not have documentation of ovarian hormonal failure must have a serum follicle stimulating hormone (FSH) level at screening within the post-menopausal range based on the Central Laboratory reference range

Key Exclusion Criteria:

* A new acquired immunodeficiency syndrome (AIDS)-defining condition diagnosed within the 30 days prior to screening
* Hepatitis B surface antigen position
* Hepatitis C antibody positive
* Participants experiencing decompensated cirrhosis
* Females who are breastfeeding
* Positive serum pregnancy test
* Have an implanted defibrillator or pacemaker
* Current alcohol or substance use judged by the Investigator to potentially interfere with subject study compliance
* History of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with dosing requirements
* Participation in any other clinical trial without prior approval from the sponsor is prohibited while participating in this trial
* Participants receiving ongoing therapy with drugs not to be used with elvitegravir (EVG), COBI, FTC, TDF, ATV, RTV, EFV, and TAF or participants with any known allergies to the excipients of E/C/F/TDF, E/C/F/TAF, EFV/FTC/TDF, ATV, COBI, RTV, or FTC/TDF

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1443 (Actual)
Dates: Start 2013-03-27 (Actual); Primary Completion 2015-03-16 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (167):
- United States (91):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Southwest Center for HIV/AIDS, Phoenix, Arizona
  - Spectrum Medical Group, Phoenix, Arizona
  - Health for Life Clinic PLLC, Little Rock, Arkansas
  - AHF Research Center, Beverly Hills, California
  - Michael Keith Wensley, MD, Inc., A Medical Corporation, Costa Mesa, California
  - Living Hope Clinical Foundation, Long Beach, California
  - Kaiser Permanente, Los Angeles, California
  - Jeffrey Goodman Special Care Clinic, Los Angeles, California
  - Peter J Ruane, MD, Inc, Los Angeles, California
  - Anthony Mills MD Inc, Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - Alameda County Medical Center, Oakland, California
  - East Bay AIDS Center, Oakland, California
  - Stanford University, Palo Alto, California
  - University of California, Davis Medical Center, Sacramento, California
  - Kaiser Permanente Medical Group, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Metropolis Medical Group, San Francisco, California
  - Kaiser Permanente Medical Center, Clinical Trials Unit, San Francisco, California
  - Kaiser Permanente Hospital, San Leandro, California
  - Apex Research LLC, Denver, Colorado
  - Greenwich Hospital, Greenwich, Connecticut
  - Yale University HIV Clinical Trials Program, New Haven, Connecticut
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Broward Health/Comprehensive Care Center, Fort Lauderdale, Florida
  - Gary J. Richmond,M.D.,P.A., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - The Kinder Medical Group, Miami, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - IDOCF/ Value Health MD, LLC, Orlando, Florida
  - University of South Florida HIV Clinical Research Unit / Hillsborough County Health Department, Tampa, Florida
  - Infectious Disease Research Institute Inc., Tampa, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Atlanta ID Group, PC, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - University of Hawaii - Hawaii Center for AIDS, Honolulu, Hawaii
  - Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - NorthStar Medical Center, Chicago, Illinois
  - Community Research Initiative of New England, Boston, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Baystate Infectious Diseases Clinical Research, Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Central West Clinical Research, St Louis, Missouri
  - Saint Louis University, St Louis, Missouri
  - Southampton Healthcare, St Louis, Missouri
  - ID Care, Hillsborough, New Jersey
  - Saint Michaels Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - SouthWest CARE Center, Santa Fe, New Mexico
  - Upstate ID Association, Albany, New York
  - Albany Medical College, Albany, New York
  - New York Hospital Queens, Flushing, New York
  - North Shore University Hospital, Divison of Infectious Diseases, Manhasset, New York
  - Greiger Clinic, Mount Vernon, New York
  - Beth Israel Medical Center- Division of Infectious Diseases, New York, New York
  - Chelsea Village Medical, PC, New York, New York
  - Ricky K. Hsu, MD, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center - AIDS Center, The Bronx, New York
  - University of NC AIDS Clinical Trials Unit, Chapel Hill, North Carolina
  - Carolinas Medical Center-Myers Park, Charlotte, North Carolina
  - Duke University Health System, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Summa Health System, Akron, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - AIDS Arms, Inc./ Peabody Health Center, Dallas, Texas
  - Southwest Infectious Disease Clinical Research, Inc., Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Garcia's Family Health Group, Harlingen, Texas
  - Therapeutic Concepts, P.A., Houston, Texas
  - Gordon E. Crofoot MD PA, Houston, Texas
  - Research Access Network, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Clinical Alliance for Research & Education, Infectious Diseases (CARE-ID), Annandale, Virginia
  - Peter Shalit, M.D., Seattle, Washington
  - Premier Clinical Research, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - East Sydney Doctors, Darlinghurst, New South Wales
  - Holdsworth House Medical practice, Darlinghurst, New South Wales
  - St Vincent's Hospital, Sydney, Darlinghurst, New South Wales
  - Taylor Square Private Clinic, Darlinghurst, New South Wales
  - Albion Street Centre, Surry Hills, New South Wales
  - Melbourne Sexual Health Clinic, Carlton, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Northside Clinic, Melbourne, Victoria
  - Prahran Market Clinic, South Yarra, Victoria
- Austria (3):
  - Medizinische Universität Graz, Graz
  - Medizinische Universitat Wien, Vienna
  - SMZ Baumgartner Hoehe - Otto-Wagner-Spital, Vienna
- Belgium (2):
  - CHU Saint-Pierre University Hospital, Brussels
  - Hôpital Universitaire Erasme - ULB, Ghent
- Brazil (4):
  - Instituto De Pesquisa Clinica Evandro Chagas - Fundação Oswaldo Cruz, Rio de Janeiro
  - Faculdade de Medicina do ABC, Santo André
  - São Paulo Secretaria da Saúde - Instituto De Infectologia Emilio Ribas, São Paulo
  - São Paulo Secretaria da Saúde - Centro de Referência e Treinamento em DST/AIDS, São Paulo
- Canada (10):
  - Ubc Downtown I.D. Clinic, Vancouver, British Columbia
  - Winnipeg Regional Health Authority - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Maple Leaf Research, Toronto, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario
  - Clinique medicale l'Actuel, Montreal, Quebec
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
  - McGill University Health Centre (MUHC) - Montral Chest Institute, Montreal, Quebec
  - Clinique OPUS, Montreal, Quebec
- Epidemiklinikken 5112, Rigshospitalet, Copenhagen, Denmark
- Instituto Dominicano de Estudios Virologicos - IDEV, Santo Domingo, Dominican Republic
- France (7):
  - Hôpital de La Croix Rousse, Lyon
  - CHU Hotel Dieu, Nantes
  - Archet 1 CHU de Nice - 6ème Niveau, Nice
  - Hôpital Saint Louis, Paris
  - Hopital Saint Antoine, Paris
  - Bichat Hospital, Paris
  - Centre Hospitalier de Tourcoing, Tourcoing
- Germany (10):
  - EPIMED GmbH, Berlin
  - University of Bonn, Bonn
  - University of Cologne, Department of Internal Medicine, Cologne
  - Center for HIV and Hepatogastroenterology, Düsseldorf
  - Infektio Research GmbH / Infektiologikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - ICH Study Center Hamburg, Hamburg
  - University Medical Center Hamburg-Eppendorf, Infectious Diseases Unit, Hamburg
  - MUC Research GmbH, München
- Italy (4):
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Azienda Ospedaliera Luigi Sacco 1° Divisione Malattie Infettive, Milan
  - Istituto Nazionale Malattie Infettive "Lazzaro Spallanzani" IRCCS, Rome
  - Comprensorio Amedeo Di Savoia Birago Di Vische, Torino
- Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Mexico
- Netherlands (2):
  - Onze Lieve Vrouwe Gasthuis, Afdeling Infectieziekten, Amsterdam
  - Erasmus MC, Rotterdam
- Portugal (2):
  - Hospital de Santa Maria, Lisbon
  - Servico De Doencas Infecciosas - Hospital De Sao Joao, Porto
- Puerto Rico (3):
  - Clinical Research Puerto Rico, San Juan, PR
  - HOPE Clinical Research, San Juan, Pr
  - VA Caribbean Healthcare System, San Juan, Pr
- Spain (3):
  - Hospital Universitari De Bellvitge, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen del Rocio, Seville
- Södersjukhuset, Stockholm, Sweden
- Switzerland (3):
  - Universitätsklinik für Infektiologie, Universitätsspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - University Hospital of Zurich, Zurich
- Thailand (5):
  - HIV-NAT, Thai Red Cross AIDS Research Center and Faculty of Medicine Chulalongkorn University, Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok
  - Siriraj HospitalDepartment of Preventive and Social Medicine, Faculty of Medicine, Bangkok
  - Maharaj Nakorn Chiang Mai University, Faculty of Medicine, Department of Medicine, Chiang Mai
  - Khon Kaen University, Khon Kaen
- United Kingdom (5):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Barts and the London NHS Trust, London
  - Chelsea and Westminster Hospital Foundation Trust, London
  - Courtyard Clinic, St. Georges Hospital, London
  - North Manchester General Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Mills A, Arribas JR, Andrade-Villanueva J, DiPerri G, Van Lunzen J, Koenig E, Elion R, Cavassini M, Madruga JV, Brunetta J, Shamblaw D, DeJesus E, Orkin C, Wohl DA, Brar I, Stephens JL, Girard PM, Huhn G, Plummer A, Liu YP, Cheng AK, McCallister S; GS-US-292-0109 team. Switching from tenofovir disoproxil fumarate to tenofovir alafenamide in antiretroviral regimens for virologically suppressed adults with HIV-1 infection: a randomised, active-controlled, multicentre, open-label, phase 3, non-inferiority study. Lancet Infect Dis. 2016 Jan;16(1):43-52. doi: 10.1016/S1473-3099(15)00348-5. Epub 2015 Nov 2. PMID 26538525
- [Result] Orkin C, DeJesus E, Ramgopal M, Crofoot G, Ruane P, LaMarca A, Mills A, Vandercam B, de Wet J, Rockstroh J, Lazzarin A, Rijnders B, Podzamczer D, Thalme A, Stoeckle M, Porter D, Liu HC, Cheng A, Quirk E, SenGupta D, Cao H. Switching from tenofovir disoproxil fumarate to tenofovir alafenamide coformulated with rilpivirine and emtricitabine in virally suppressed adults with HIV-1 infection: a randomised, double-blind, multicentre, phase 3b, non-inferiority study. Lancet HIV. 2017 May;4(5):e195-e204. doi: 10.1016/S2352-3018(17)30031-0. Epub 2017 Mar 2. PMID 28259777
- [Result] Brown T, Yin MT, Gupta S, Katlama C, et al. Switching from TDF to TAF in HIV-infected adults with low BMD: a pooled analysis. 24th Annual Conference on Retroviruses and Opportunistic Infections (CROI) - CROI Foundation 2017; poster presentation: abstract #683.
- [Result] Podzamczer D, Viciana P, Rijnders B, Shalit P, et al. Switching from Tenofovir disoproxil fumarate to tenofovir alafenamide in patients with high risk for chronic kidney disease. 8th National Congress of the AIDS Study Group (GESIDA) and Spanish Society of Infectious Diseases and Clinical Microbiology (SEIMC) held jointly with the 9th Teacher Meeting of AIDS Research Network 2016; poster presentation: abstract #P-188.
- [Result] Orkin C, Rjinders B, Stephan C, McKellar M, et al. Switching from boosted atazanavir (ATV) plus FTC/TDF to a TAF-based single tablet regimen (STR): Week 48 data in virologically suppressed adults. Annual Conference of the British Association for Sexual Health and HIV (BASHH) 2016; poster presentation: abstract # P045.
- [Result] Mills A, Andrade J, Koenig E, et al. Switching from a tenofovir disoproxil fumarate (TDF)-based regimen to a tenofovir alafenamide (TAF)-based regimen: data in virologically suppressed adults through 48 weeks of treatment. 13th Congress for Infectious Diseases and Tropical Medicine (KIT) 2016; poster presentation: abstract #eP-038.
- [Result] Overton ET, Shalit P, Crofoot G, Benson P, et al. Switch from TDF regimens to E/C/F/TAF is associated with improved bone mineral density (BMD), decreased serum PTH and decreased bone turnover biomarkers. 56th Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC) held Jointly with the 2016 Annual Meeting on Microbe - American Society for Microbiology (ASM) 2016; poster presentation: abstract #PW-027.
- [Result] Huhn G, Rijnders B, Thompson M, Tebas P, et al. Switching from TDF to TAF in patients with high risk for CKD. 56th Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC) held Jointly with the 2016 Annual Meeting on Microbe - American Society for Microbiology (ASM) 2016; oral presentation: https://www.natap.org/2016/HIV/062116_01.htm.
- [Result] Abram M, Margot NA, Cox S, Ram RR, et al. Pooled week-48 analysis of HIV-1 drug resistance in E/C/F/TAF (Genvoya) phase 3 studies. 23rd Annual Conference on Retroviruses and Opportunistic Infections (CROI) - CROI Foundation 2016, poster presentation: abstract #496.
- [Result] Abram M, Margot NA, Cox S, Ram RR, et al. Pooled week-48 analysis of HIV-1 drug resistance in E/C/F/TAF (Genvoya) phase 3 studies. 25th International HIV Drug Resistance Workshop - Informed Horizons, LLC 2016; poster presentation: abstract #33.
- [Result] Mills A, Andrade J, Di Perri G, Van Lunzen J, et al. Switching from a tenofovir disoproxil fumarate (TDF)-based regimen to a tenofovir alafenamide (TAF)-based regimen: data in virologically suppressed adults through 48 weeks of treatment. 8th Biennial Conference on HIV Pathogenesis and Treatment and Prevention of the International AIDS Society (IAS) 2015; oral presentation: abstract #TUAB0102.
- [Result] Shamblaw D, Van Lunzen J, Orkin C, Bloch M, eta al. Switching from Atripla (ATR) to a tenofovir alafenamide (TAF)-based single tablet regimen: week 48 data in virologically suppressed adults. 55th Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC) 2015; oral presentation; https://natap.org/2015/ICAAC/ICAAC_13.htm.
- [Result] Thompson M, Morales-Ramirez J, Mcdonald C, Rachlis A, et al. Switching from a tenofovir disoproxil fumarate (TDF) to a tenofovir alafenamide (TAF)-based single tablet regimen (STR): Week 48 data in HIV-1 infected virologically suppressed adults. Spring Conference of the Society for Healthcare Epidemiology of America (SHEA) 2015; oral presentation: abstract #725.
- [Result] Rijnders B, Stephan C, Lazzarin A, Squires K, et al. Switching from ritonavir or cobicistat boosted atazanavir (ATV) plus emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) to a tenofovir alafenamide (TAF)-based single tablet regimen (STR): week 48 data in virologically suppressed adults. 15th European AIDS Conference (EACS) and 17th International Workshop on Co-morbidities and Adverse Drug Reactions in HIV 2015; poster presentation: abstract #577.
- [Result] Lutz T, Benson P, Goffard J-C, Haubrich R, et al. Patient reported outcomes (PRO) over 48 weeks in a randomized, open-label trial of patients with HIV switching to coformulated elvitegravir, cobicistat, emtricitabine, and tenofovir alafenamide (E/C/F/TAF). 15th European AIDS Conference (EACS) and 17th International Workshop on Co-morbidities and Adverse Drug Reactions in HIV 2015; poster presentation: abstract #324.
- [Result] Viciana P, Mills A, Andrade J, Diperri G, et al. Switching from a tenofovir disoproxil fumarate (TDF)-based regimen to a tenofovir alafenamide (TAF)-based regimen: data in virologically suppressed adults through 48 weeks of treatment. 7th National Congress of the AIDS Study Group (GESIDA) and Spanish Society of Infectious Diseases and Clinical Microbiology (SEIMC) held jointly with the 8th Teacher Meeting of AIDS Research Network 2015; oral presentation: abstract #PO-08.
- [Result] Mills A, Andrade-Villanueva J, DiPerri G, Van Luzen J, et al. Switching from a tenofovir disoproxil fumarate (TDF)-based regimen to a tenofovir alafenamide (TAF)-based regimen: Data in virologically suppressed adults through 48 weeks of treatment. 8th Annual International AIDS Society meeting 2015; oral presentation: abstract #839.
- [Result] Thompson M, Brar I, Brinson C, Creticos C, et al. Tenofovir alafenamide vs tenofovir DF in women: pooled analysis of 7 clinical trials. Annual Meeting of the American Pharmacists Association (APhA) - Virtual 2020; poster presentation: abstract #209.
- [Result] Stellbrink H, Gandhi-Patel B, Zhong L, Das M, et al. Safety and efficacy of switching from tenofovir disoproxil fumarate to tenofovir alafenamide in people with HIV aged 50 years and older. Annual Meeting of the American Pharmacists Association (APhA) - Virtual 2020; poster presentation: abstract #205.
- [Result] Stellbrink H-J, Post FA, Podzamczer D, Arribas J, et al. Safety and efficacy of switching from tenofovir disoproxil fumarate to tenofovir alafenamide in people with HIV aged 50 years and older. 15th Congress on Infectious Diseases and Tropical Medicine - German Society for Infectious Diseases (DPID) held jointly with the 29th Annual Meeting of the German Society for Pediatric Infectiology (DGPI) 2020; poster presentation: abstract #A-343.
- [Result] Gupta SK, Post FA, Arribas JR, Eron JJ Jr, Wohl DA, Clarke AE, Sax PE, Stellbrink HJ, Esser S, Pozniak AL, Podzamczer D, Waters L, Orkin C, Rockstroh JK, Mudrikova T, Negredo E, Elion RA, Guo S, Zhong L, Carter C, Martin H, Brainard D, SenGupta D, Das M. Renal safety of tenofovir alafenamide vs. tenofovir disoproxil fumarate: a pooled analysis of 26 clinical trials. AIDS. 2019 Jul 15;33(9):1455-1465. doi: 10.1097/QAD.0000000000002223. PMID 30932951
- [Result] Hermansson L, Yilmaz A, Price RW, Nilsson S, McCallister S, Makadzange T, Das M, Zetterberg H, Blennow K, Gisslen M. Plasma concentration of neurofilament light chain protein decreases after switching from tenofovir disoproxil fumarate to tenofovir alafenamide fumarate. PLoS One. 2019 Dec 11;14(12):e0226276. doi: 10.1371/journal.pone.0226276. eCollection 2019. PMID 31826005
- [Result] Stellbrink H-J, Post FA, Podzamczer D, Arribas J, et al. Safety and efficacy of switching from tenofovir disoproxil fumarate to tenofovir alafenamide in people with HIV aged 50 years and older. 17th European AIDS Conference of the European AIDS Clinical Society (EACS) 2019; poster presentation: abstract #PE9-50.
- [Result] Pepperrell T, Hughes S, Gotham D, Pozniak A, et al. Tenofovir alafenamide versus tenofovir disoproxil fumarate - is there a true difference in safety? 17th European AIDS Conference of the European AIDS Clinical Society (EACS) 2019; poster presentation: abstract #PE3-8.
- [Result] Thompson M, Brar I, Brinson C, Creticos C, et al. Tenofovir alafenamide vs. tenofovir DF in women: pooled analysis of 7 clinical trials. 9th Edition International Workshop on HIV and Women - Virology Education 2019; poster presentation: abstract #21.
- [Result] Dejesus E, Federico Andrade Villanueva J, Ramon Arribas Lopez J, Brinson C, et al. Tenofovir alafenamide (TAF) versus tenofovir disoproxil fumarate (TDF) in hispanic/latinx and black participants: efficacy, bone and renal safety results from a pooled analysis of 7 clinical trials. IDWeek Meeting of the Infectious Diseases Society of America (IDSA) 2019; poster presentation: abstract #318.
- [Result] Walmsley S, Andany N, Brar I, Brinson C, et al. Tenofovir alafenamide VS tenofovir DF in women: pooled analysis of 7 clinical trials. 28th Annual Canadian Conference on HIV/AIDS Research - Canadian Association for HIV Research (CAHR) 2019; poster presentation: abstract #CSP9.04.
- [Result] Kim YS, Oka S, Chetchotisakd P, Clarke A, Supparatpinyo K, Avihingsanon A, Ratanasuwan W, Kiertiburanakul S, Ruxrungtham K, Yang S, Guo S, Liu Y, Das M, Tran D, McColl D, Corales R, Nguyen C, Piontkowsky D. Efficacy and safety of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide in Asian participants with human immunodeficiency virus 1 infection: A sub-analysis of phase 3 clinical trials. HIV Res Clin Pract. 2019 Jun;20(3):73-81. doi: 10.1080/15284336.2019.1589232. Epub 2019 Jul 8. PMID 31303140
- [Result] Hermansson L, Price RW, Yilmaz A, Nilsson S, et al. Effect on plasma NFL, a marker or neuronal injury, after switching from TDF to TAF. Annual Conference on Retroviruses and Opportunistic Infections (CROI) - CROI Foundation 2019; oral presentation: abstract #127.
- [Result] Thompson M, Brar I, Brinson C, Creticos C, et al. Tenofovir alafenamide VS tenofovir DF in women: pooled analysis of 7 clinical trials. Annual Conference on Retroviruses and Opportunistic Infections (CROI) - CROI Foundation 2019; poster presentation: abstract #519.
- [Result] Orkin C, Castelli F, Yazdanpanah Y, Rockstroh J, et al. Cardiovascular disease risk assessments and fasting lipid changes in virologically suppressed patients randomized to switch to tenofovir alafenamide versus continuing tenofovir disoproxil fumarate. 22nd International AIDS Conference - International AIDS Society 2018; poster presentation: abstract #TUPEB104.
- [Result] Brown TT, Yin MT, Gupta SK, Short WR, et al. Combined effects of bisphosphonates & TDF->TAF switch in HIV+ adults with low BMD. Annual Conference on Retroviruses and Opportunistic Infections (CROI) - CROI Foundation 2018; poster presentation: abstract #724.
- [Result] DeJesus E, Haas B, Segal-Maurer S, Ramgopal MN, Mills A, Margot N, Liu YP, Makadzange T, McCallister S. Superior Efficacy and Improved Renal and Bone Safety After Switching from a Tenofovir Disoproxil Fumarate- to a Tenofovir Alafenamide-Based Regimen Through 96 Weeks of Treatment. AIDS Res Hum Retroviruses. 2018 Apr;34(4):337-342. doi: 10.1089/AID.2017.0203. Epub 2018 Mar 20. PMID 29368537
- [Result] Goldstein D, Ward D, Brinson C, Crofoot G, et al. Week 96 efficacy and safety of tenofovir alafenamide (TAF) versus tenofovir disoproxil fumarate (TDF) in older, HIV-Infected virologically-suppressed adults. Annual Meeting of the American Geriatrics Society (AGS) 2017; poster presentation: abstract #A90.
- [Result] Ward D, Thompson M, Goldstein D, Brinson C, et al. Week 96 efficacy and safety of tenofovir alafenamide (TAF) versus tenofovir disoproxil fumarate (TDF) in older, HIV-infected treatment-naïve adults. Annual Meeting of the American Geriatrics Society (AGS) 2017; poster presentation: abstract #A91.
- [Result] Choe S, Podzamvzer D, Tashima K, McNicholl I, and McCallister S. Utilizing phase 3 clinical trial data to assess adverse event (AE) frequency of a potentially interacting medication (PIM) amlodipine with elvitegravir/cobicistat (EVG/COBI). Midyear Clinical Meeting of the American Society of Health-System Pharmacists (ASHP) 2017; poster presentation: abstract #7-068.
- [Result] Yin M, Gupta S, Nguyen-Cleary T, Mora M, and Das M. Switching from TDF to TAF in HIV-infected adults with low BMD: A pooled analysis. Congress on HIV and Hepatitis in the Americas - ViiV Healthcare UK Limited 2017; poster presentation: abstract #P021.
- [Result] Podzamczer D, Tashima K, Daar E, McGowan J, et al. Utilizing phase 3 clinical trial data to assess adverse event (AE) frequency of a potentially interacting medication (PIM) amlodipine with elvitegravir/cobicistat (EVG/COBI). International Congress of Drug Therapy in HIV Infection - International AIDS Society 2016; poster presentation: abstract #P314.
- [Result] Dejesus E, Haas B, Segal-Maurer S, Ramgopal M, et al. Superior efficacy and improved renal and bone safety after switching from a tenofovir disoproxil fumarate (TDF) regimen to a tenofovir alafenamide (TAF) based regimen through 96 weeks (W96) of treatment. 56th Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC) held Jointly with the 2016 Annual Meeting on Microbe - American Society for Microbiology (ASM) 2016; poster presentation: abstract # LB-087.
- [Result] Viciana P, Rijnders B, Shalit P, Liu Y et al. Cambio desde TDF a TAF en pacientes en alto riesgo de erc. 18th Congress of the Andalusian Society of Infectious Diseases (SAID) 2016; poster presentation: abstract #P-070.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Dominican Republic, Puerto Rico, North America, South America, Europe, Australia, and Asia. The first participant was screened on 27 March 2013. The last study visit occurred on 01 April 2020.
Pre-assignment Details: 1559 participants were screened.
Groups:
- E/C/F/TAF: Randomized Phase: Elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) (150/150/200/10 mg) fixed-dose combination (FDC) tablet administered once daily for up to 96 weeks.
  Extension Phase: After completing 96 weeks of randomized treatment, all participants were given the opportunity to receive open-label E/C/F/TAF until it became commercially available, or until Gilead elected to terminate the development of E/C/F/TAF.
- Stay on Baseline Treatment Regimen (SBR): Randomized Phase: Participants stayed on their baseline emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF)-containing regimen (E/C/F/TDF; efavirenz (EFV)/FTC/TDF; ritonavir (RTV)-boosted atazanavir (ATV)+FTC/TDF; or cobicistat (COBI-boosted ATV+FTC/TDF)) administered according to prescribing information for up to 96 weeks.
  Extension Phase: After completing 96 weeks of randomized treatment (SBR), all participants were given the opportunity to receive open-label E/C/F/TAF until it became commercially available, or until Gilead elected to terminate the development of E/C/F/TAF.
Period: Randomized Treatment Phase-Up to Week 96
Arm/Group | E/C/F/TAF | Stay on Baseline Treatment Regimen (SBR)
Started | 963 | 480
Completed | 914 | 445
Not Completed | 49 | 35
Not completed — Withdrew Consent | 11 | 17
Not completed — Lost to Follow-up | 10 | 9
Not completed — Investigator's Discretion | 11 | 2
Not completed — Adverse Event | 7 | 4
Not completed — Death | 4 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Participants randomized and never treated | 4 | 3
Period: Extension Treatment Phase- After Week 96
Arm/Group | E/C/F/TAF | Stay on Baseline Treatment Regimen (SBR)
Started | 905 (9 participants who completed the Randomized Treatment Phase did not continue in the Extension E/C/F/TAF Treatment Phase.) | 424 (21 participants who completed the Randomized Treatment Phase did not continue in the Extension E/C/F/TAF Treatment Phase.)
Completed | 854 | 398
Not Completed | 51 | 26
Not completed — Investigator's Discretion | 31 | 15
Not completed — Lost to Follow-up | 13 | 9
Not completed — Withdrew Consent | 5 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who were randomized and received at least one dose of study drug.
Groups:
- E/C/F/TAF: Randomized Phase: Elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF)(150/150/200/10 mg) fixed-dose combination (FDC) tablet administered once daily for up to 96 weeks.
  Extension Phase: After completing 96 weeks of randomized treatment, all participants were given the opportunity to receive open-label E/C/F/TAF until it became commercially available, or until Gilead elected to terminate the development of E/C/F/TAF.
- Total: Total of all reporting groups
Arm/Group | E/C/F/TAF | Stay on Baseline Treatment Regimen (SBR) | Total
Number analyzed (Participants) | 959 | 477 | 1436
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41 (10.1) | 41 (10.1) | 41 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 50 | 153
  Male | 856 | 427 | 1283
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 5 | 2 | 7
  Race: Asian | 59 | 35 | 94
  Race: Black | 169 | 102 | 271
  Race: Native Hawaiian or Pacific Islander | 6 | 1 | 7
  Race: White | 651 | 314 | 965
  Race: Local regulators did not allow collection of race or ethnicity information | 2 | 1 | 3
  Race: Other | 67 | 22 | 89
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 248 | 82 | 330
  Ethnicity: Not Hispanic or Latino | 709 | 392 | 1101
  Ethnicity: Local regulators did not allow collection of race or ethnicity information | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 648 | 316 | 964
  United Kingdom | 14 | 8 | 22
  Thailand | 35 | 21 | 56
  Portugal | 8 | 2 | 10
  Switzerland | 5 | 4 | 9
  Spain | 5 | 3 | 8
  Canada | 51 | 27 | 78
  Austria | 16 | 8 | 24
  Netherlands | 2 | 3 | 5
  Sweden | 1 | 0 | 1
  Belgium | 14 | 8 | 22
  Brazil | 14 | 5 | 19
  Denmark | 1 | 2 | 3
  Dominican Republic | 29 | 13 | 42
  Italy | 13 | 6 | 19
  Mexico | 19 | 6 | 25
  Australia | 38 | 22 | 60
  France | 12 | 12 | 24
  Germany | 34 | 11 | 45
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 943 | 466 | 1409
  ≥ 50 copies/mL | 16 | 11 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Full Analysis Set included participants who were randomized and received at least 1 dose of study drug.
  New Drug Application (NDA Data Cut) = participants through the data cut for the E/C/F/TAF NDA; All Participants = participants through the Week 48 Data Cut.
Measure: Number; unit: percentage of participants
Groups:
- E/C/F/TAF: Elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) (150/150/200/10 mg) FDC tablet administered once daily for up to 96 weeks in the Randomized Phase.
- Stay on Baseline Treatment Regimen (SBR): Participants stayed on their baseline emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF)-containing regimen (E/C/F/TDF; efavirenz (EFV)/FTC/TDF; ritonavir (RTV)-boosted atazanavir (ATV)+FTC/TDF; or cobicistat (COBI-boosted ATV+FTC/TDF)) administered according to prescribing information for up to 96 weeks in the Randomized Phase.
Arm/Group | E/C/F/TAF | Stay on Baseline Treatment Regimen (SBR)
Number analyzed (Participants) | 959 | 477
percentage of participants
  NDA Data Cut: number analyzed (Participants) | 799 | 397
  NDA Data Cut | 95.6 | 92.9
  All Participants | 97.2 | 93.1
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); NDA Data Cut; Test type: Non-Inferiority or Equivalence — Null hypothesis: the E/C/F/TAF group was at least 12% worse than the Stay on Baseline Regimen group; alternative hypothesis: the E/C/F/TAF group was less than 12% worse than the in Stay on Baseline Regimen group; p = 0.051, Cochran-Mantel-Haenszel — The p-value for the superiority test used a 2-sided Cochran-Mantel-Haenszel (CMH) test, stratified by prior treatment regimen; Difference in percentages = 2.7, 95.01% CI 2-sided [-0.3 to 5.6] — The difference in percentages and its 95.01% confidence interval (CI) were calculated based on the Mantel-Haenszel (MH) proportion adjusted by the prior treatment regimen
Statistical Analysis 2: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); All Participants; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentages = 4.1, 95% CI 2-sided [1.6 to 6.7] — The difference in percentages and its 95% confidence interval (CI) were calculated based on the Mantel-Haenszel (MH) proportion adjusted by the prior treatment regimen

2. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 48
Description: Hip BMD was assessed by dual energy x-ray absorptiometry (DXA) scan. BMD is calculated as grams per square centimeter (g/cm^2); the mean (SD) percentage change is presented.
Time Frame: Baseline; Week 48
Population: Participants in the Hip DXA Analysis Set (participants who received ≥ 1 dose of study drug and had nonmissing baseline hip BMD) with available data were analyzed.
  NDA Data Cut = participants through the data cut for the E/C/F/TAF NDA; All Participants = participants through the Week 48 Data Cut.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | E/C/F/TAF | Stay on Baseline Treatment Regimen (SBR)
Number analyzed (Participants) | 902 | 452
percentage change
  NDA Data Cut: number analyzed (Participants) | 733 | 350
  NDA Data Cut | 1.949 (2.9956) | -0.136 (2.9890)
  All Participants: number analyzed (Participants) | 869 | 428
  All Participants | 1.468 (2.7136) | -0.340 (2.8280)
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); NDA Data Cut; Test type: Superiority or Other; p < 0.001, ANOVA — P-value was from the analysis of variance (ANOVA) model including study treatment and prior treatment regimen as fixed effects; Difference in least square means = 2.078, 95% CI 2-sided [1.697 to 2.459] — Difference in least squares means (LSM) and its 95% CI were from the ANOVA model including treatment and prior treatment regimen as fixed effects
Statistical Analysis 2: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); All Participants; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least square means = 1.807, 95% CI 2-sided [1.488 to 2.126] — Difference in least squares means and its 95% CI were from the ANOVA model including treatment and prior treatment regimen as fixed effects

3. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 48
Description: Spine BMD was assessed by DXA scan. BMD is calculated as g/cm^2; the mean (SD) percentage change is presented.
Time Frame: Baseline; Week 48
Population: Participants in the Spine DXA Analysis Set (participants who received ≥ 1 dose of study drug and had nonmissing baseline spine BMD) with available data were analyzed.
  NDA Data Cut = participants through the data cut for the E/C/F/TAF NDA; All Participants = participants through the Week 48 Data Cut.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | E/C/F/TAF | Stay on Baseline Treatment Regimen (SBR)
Number analyzed (Participants) | 912 | 457
percentage change
  NDA Data Cut: number analyzed (Participants) | 742 | 356
  NDA Data Cut | 1.861 (3.0889) | -0.110 (3.7415)
  All Participants: number analyzed (Participants) | 881 | 436
  All Participants | 1.557 (3.8441) | -0.443 (4.1387)
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); NDA Data Cut; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least square means = 1.970, 95% CI 2-sided [1.551 to 2.390] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); All Participants; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least square means = 2.000, 95% CI 2-sided [1.549 to 2.452] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Safety Analysis Set (randomized participants who received ≥ 1 dose of study drug) excluding participants with prior treatment of EFV/FTC/TDF.
  NDA Data Cut = participants through the data cut for the E/C/F/TAF NDA; All Participants = participants through the Week 48 Data Cut
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | E/C/F/TAF | Stay on Baseline Treatment Regimen (SBR)
Number analyzed (Participants) | 708 | 352
mg/dL
  NDA Data Cut: number analyzed (Participants) | 545 | 266
  NDA Data Cut | -0.01 (0.117) | 0.04 (0.123)
  All Participants: number analyzed (Participants) | 696 | 330
  All Participants | 0.00 (0.115) | 0.03 (0.105)
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); NDA Data Cut; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was from analysis of covariance (ANCOVA) model including study treatment and prior treatment as fixed effects and baseline serum creatinine as a covariate; Difference in least square means = -0.05, 95% CI 2-sided [-0.07 to -0.03] — Difference in least squares means (LSM) and its 95% CI were from the analysis of covariance (ANCOVA) model including study treatment and prior treatment regimen as fixed effects and baseline serum creatinine as a covariate
Statistical Analysis 2: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); All Participants; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Difference in least square means = -0.04, 95% CI 2-sided [-0.05 to -0.02] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in the Overall EFV-related Symptom Assessment Score at Week 48
Description: The mean (SD) change of the overall EFV-related symptom assessment score is presented. The overall symptom score (ranging from 0 to 20) is the sum of the individual symptom scores ranging from 0 (no symptoms) to 4 (most severe symptoms) from the 5 EFV-related symptom assessments (dizziness, trouble sleeping, impaired concentration, sleepiness, and abnormal or vivid dream). A negative change from baseline indicates improvement.
  EFV-Related Symptom Analysis Set: participants who received EFV/FTC/TDF as prior treatment, received at least 1 dose of study drug, and completed EFV-related symptom assessments at the baseline visit and at least 1 postbaseline visit.
Time Frame: Baseline; Week 48
Population: Participants in EFV-Related Symptom Analysis Set with available data were analyzed.
  NDA Data Cut = participants through data cut for E/C/F/TAF NDA; All Participants = participants through Week 48 Data Cut
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | E/C/F/TAF | Stay on Baseline Treatment Regimen (SBR)
Number analyzed (Participants) | 239 | 116
units on a scale
  NDA Data Cut: number analyzed (Participants) | 210 | 96
  NDA Data Cut | -1.6 (3.06) | -0.1 (2.43)
  All Participants: number analyzed (Participants) | 224 | 101
  All Participants | -1.5 (3.06) | -0.1 (2.39)
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); NDA Data Cut; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — The P-value comparing the 2 treatment groups was from the 2-sided Wilcoxon rank sum test
Statistical Analysis 2: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); All Participants; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — The P-value comparing the 2 treatment groups was from the 2-sided Wilcoxon rank sum test

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | Stay on Baseline Treatment Regimen (SBR)
Number analyzed (Participants) | 959 | 477
percentage of participants | 92.8 | 89.1
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.017, Cochran-Mantel-Haenszel — P-value for the superiority test comparing the percentages of virologic success was from the CMH test stratified by the prior treatment regimen (STB, ATR, ATV/boosted+TVD); Difference in percentages = 3.7, 95% CI 2-sided [0.4 to 7.0] — The difference in percentages of virologic success and its 95% CI were calculated based on the MH proportion adjusted by the prior treatment regimen

7. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 20 Copies/mL at Week 48
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed. NDA Data Cut = participants through the data cut for the E/C/F/TAF NDA; All Participants = participants through the Week 48 Data Cut.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | Stay on Baseline Treatment Regimen (SBR)
Number analyzed (Participants) | 959 | 477
percentage of participants
  NDA Data Cut: number analyzed (Participants) | 799 | 397
  NDA Data Cut | 92.2 | 90.4
  All Participants | 93.5 | 90.4
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); NDA Data Cut; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.29, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 1]; Difference in percentages = 1.8, 95% CI 2-sided [-1.7 to 5.3] — Difference in percentages of virologic success and its 95% CI were calculated based on the MH proportion adjusted by the prior treatment regimen
Statistical Analysis 2: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); All Participants; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.031, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 1]; Difference in percentages = 3.2, 95% CI 2-sided [0.1 to 6.3] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 20 Copies/mL at Week 96
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | Stay on Baseline Treatment Regimen (SBR)
Number analyzed (Participants) | 959 | 477
percentage of participants | 90.6 | 85.3
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 1]; Difference in percentages = 5.3, 95% CI 2-sided [1.6 to 9.0] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Change From Baseline in Cluster Determinant 4 (CD4) Cell Count at Week 48
Description: The analysis of CD4 cell count included values up to 1 day after the last dose date of randomized study drug.The change from baseline in CD4 cell count for the full analysis set was based on observed data (ie, Missing = Excluded) for the total and by the prior treatment regimen.
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed. NDA Data Cut = participants through the data cut for the E/C/F/TAF NDA; All Participants = participants through the Week 48 Data Cut.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | E/C/F/TAF | Stay on Baseline Treatment Regimen (SBR)
Number analyzed (Participants) | 959 | 477
cells/uL
  Baseline (NDA Data Cut): number analyzed (Participants) | 799 | 397
  Baseline (NDA Data Cut) | 712 (267.9) | 690 (251.4)
  Change at Week 48 (NDA Data Cut): number analyzed (Participants) | 773 | 374
  Change at Week 48 (NDA Data Cut) | 33 (166.6) | 27 (160.2)
  Baseline (All Participants) | 701 (261.8) | 689 (248.0)
  Change at Week 48 (All Participants): number analyzed (Participants) | 937 | 449
  Change at Week 48 (All Participants) | 35 (164.6) | 24 (156.1)
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); NDA Data Cut: Change at Week 48; Test type: Superiority; p = 0.56, ANOVA — P-values were from the analysis of variance (ANOVA) model including treatment (E/C/F/TAF vs. SBR) and prior treatment regimen (STB, ATR, ATV/boosted+TVD) as fixed effects; Difference in least squares means = 6, 95% CI 2-sided [-14 to 26] — Difference in least squares means (Diff in LSM), and its 95% CI were from the analysis of variance (ANOVA) model including treatment (E/C/F/TAF vs. FTC/TDF+3rd Agent) and prior treatment regimen (STB, ATR, ATV/boosted+TVD) as fixed effects
Statistical Analysis 2: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); All Participants: Change at Week 48; Test type: Superiority; p = 0.26, ANOVA — [p-value comment as in outcome 9, analysis 1]; Difference in least squares means = 11, 95% CI 2-sided [-8 to 29] — Difference in least squares means and its 95% CI were from the analysis of variance (ANOVA) model including treatment (E/C/F/TAF vs.SBR) and prior treatment regimen (STB, ATR, ATV/boosted+TVD) as fixed effects

10. Secondary Outcome: Change From Baseline in CD4 Cell Count at Weeks 96
Description: as for outcome 9
Time Frame: Baseline; Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | E/C/F/TAF | Stay on Baseline Treatment Regimen (SBR)
Number analyzed (Participants) | 959 | 477
cells/uL
  Baseline | 701 (261.8) | 689 (248.0)
  Change at Week 96: number analyzed (Participants) | 892 | 427
  Change at Week 96 | 60 (181.6) | 42 (158.0)
Statistical Analysis 1: Comparison: E/C/F/TAF vs Stay on Baseline Treatment Regimen (SBR); Test type: Superiority; p = 0.074, ANOVA — [p-value comment as in outcome 9, analysis 1]; Difference in least squares means = 18, 95% CI 2-sided [-2 to 38] — Difference in least squares means and its 95% CI were from the analysis of variance (ANOVA) model including treatment (E/C/F/TAF vs. SBR) and prior treatment regimen (STB, ATR, ATV/boosted+TVD) as fixed effects

ADVERSE EVENTS:
Time Frame: From the first dose date up to last dose date ( maximum: 307.7 weeks) plus 30 days
Description: Safety Analysis Set included participants who were randomized and received at least one dose of study drug.
  For All Cause Mortality: All Randomized Analysis Set included all participants who were randomized into the study.
Groups:
- Randomized Phase: E/C/F/TAF: Elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (Genvoya®; EVG/COBI/FTC/TAF; E/C/F/TAF) (150/150/200/10 mg) FDC tablet administered once daily for up to 96 weeks in the Randomized Phase.
- Randomized Phase: Stay on Baseline Treatment Regimen (SBR): Participants stayed on their baseline emtricitabine(FTC)/tenofovir disoproxil fumarate (TDF)-containing regimen E/C/F/TDF (Stribild®); efavirenz (EFV)/FTC/TDF (Atripla®); ritonavir (RTV)-boosted atazanavir (ATV)+FTC/TDF; or cobicistat (COBI-boosted ATV+FTC/TDF) administered according to prescribing information for up to 96 weeks in the Randomized Phase.
- Extension Phase: E/C/F/TAF From E/C/F/TAF: After completing 96 weeks of randomized treatment (E/C/F/TAF), all participants were given the opportunity to receive open-label E/C/F/TAF in the extension phase until it became commercially available, or until Gilead elected to terminate the development of E/C/F/TAF.
- Extension Phase: E/C/F/TAF From SBR: After completing 96 weeks of randomized treatment (SBR), all participants were given the opportunity to receive open-label E/C/F/TAF in the extension phase until it became commercially available, or until Gilead elected to terminate the development of E/C/F/TAF.
Arm/Group | Randomized Phase: E/C/F/TAF | Randomized Phase: Stay on Baseline Treatment Regimen (SBR) | Extension Phase: E/C/F/TAF From E/C/F/TAF | Extension Phase: E/C/F/TAF From SBR
All-Cause Mortality (participants affected / at risk) | 4/963 | 0/480 | 1/905 | 1/424
Serious Adverse Events (participants affected / at risk) | 79/959 | 39/477 | 27/905 | 22/424
Other Adverse Events (participants affected / at risk) | 620/959 | 286/477 | 298/905 | 144/424
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Phase: E/C/F/TAF (N=959) | Randomized Phase: Stay on Baseline Treatment Regimen (SBR) (N=477) | Extension Phase: E/C/F/TAF From E/C/F/TAF (N=905) | Extension Phase: E/C/F/TAF From SBR (N=424)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0 | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 2 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Sudden death (General disorders) | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0
Vascular stent occlusion (General disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0
Acute hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Appendiceal abscess (Infections and infestations) | 0 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 3 | 1 | 1 | 1
Bacterial colitis (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 2 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Gonorrhoea (Infections and infestations) | 1 | 0 | 0 | 0
H1n1 influenza (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis A (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis syphilitic (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis aseptic (Infections and infestations) | 3 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 1
Neurosyphilis (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 2 | 0 | 0
Parasitic gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Perineal infection (Infections and infestations) | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 0 | 0 | 2
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Reiter's syndrome (Infections and infestations) | 1 | 0 | 0 | 0
Scrotal infection (Infections and infestations) | 0 | 1 | 0 | 0
Secondary syphilis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 4 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0
Device breakage (Product Issues) | 0 | 0 | 0 | 1
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Substance abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 2 | 0 | 0 | 0
Suicidal behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 4 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 1 | 0
Bladder disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Fanconi syndrome acquired (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Substance use (Social circumstances) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Phase: E/C/F/TAF (N=959) | Randomized Phase: Stay on Baseline Treatment Regimen (SBR) (N=477) | Extension Phase: E/C/F/TAF From E/C/F/TAF (N=905) | Extension Phase: E/C/F/TAF From SBR (N=424)
Diarrhoea (Gastrointestinal disorders) | 109 | 51 | 40 | 22
Nausea (Gastrointestinal disorders) | 56 | 18 | 8 | 13
Pyrexia (General disorders) | 48 | 21 | 7 | 6
Bronchitis (Infections and infestations) | 69 | 26 | 17 | 13
Nasopharyngitis (Infections and infestations) | 96 | 48 | 47 | 20
Pharyngitis (Infections and infestations) | 56 | 14 | 15 | 5
Sinusitis (Infections and infestations) | 58 | 31 | 25 | 9
Syphilis (Infections and infestations) | 63 | 38 | 19 | 9
Upper respiratory tract infection (Infections and infestations) | 168 | 64 | 67 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 78 | 31 | 19 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 70 | 33 | 30 | 9
Osteopenia (Musculoskeletal and connective tissue disorders) | 67 | 25 | 28 | 13
Headache (Nervous system disorders) | 83 | 25 | 18 | 9
Depression (Psychiatric disorders) | 48 | 30 | 15 | 7
Insomnia (Psychiatric disorders) | 58 | 36 | 12 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 73 | 31 | 28 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 57 | 12 | 10 | 7

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years